CLINICAL TRIAL: NCT03246516
Title: Individual and Socio-economic Determinants of Patient Delay in Doctor Consultation in Oeso-gastric Cancers
Brief Title: Determinants of Patient Delay in Doctor Consultation in Oeso-gastric Cancers
Acronym: DELOGAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: University of Lille Nord de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015_74; 2015-A01986-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Oesophageal Carcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire (Experimental): Auto and hetero questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Auto and hetero questionnaires:
  * STAI Y B, State-Trait Anxiety Inventoriage
  * Brief COPE
  * RHHI-24, Revised Health Hardiness Inventory
  * IPQ-R, Illness Perception Questionnaire

SUMMARY:
This study evaluates the role of socioeconomic and individual factors in the onset of the first symptoms of cancer and the first consultation with a doctor (patient delay) in oeso-gastric cancer.

DETAILED DESCRIPTION:
Reducing the time between the onset of the first symptoms of cancer and the first consultation with a doctor (patient delay) is essential to improve the vital prognosis and quality of life of patients. Recent data suggest that some sociocognitive and emotional determinants may explain patient delay from a complementary point of view. The main objective of this study is to assess whether, in oeso-gastric cancer, patient delay is linked to these sociocognitive and emotional factors, in addition to previously known factors.

We intend to include in this study 300 patients with a not yet treated oeso-gastric cancer diagnosed in one of 10 health centres in the North of France region. The collected data will be analysed to underline the differences between patients who consulted a doctor earlier versus those who consulted later with a cut off at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* oesophageal, oeso-gastric junction or gastric cancer non treated cancer
* patient informed of his diagnosis
* speak fluent french

Exclusion Criteria:

* history of cancer
* psychological history
* patient under guardianship-
* fortuitous diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Time limit of first doctor consultation | baseline
  Median time between date of symptoms appearance and date of first consultation

SECONDARY OUTCOMES:
Time limit of system of care | baseline
  Median time between date of he beginning of clinical investigations and the beginning of treatment
cTNM Stage | baseline
  Stage TNM by distinguishing the early stages (I, II) vs. (III, IV)
clinical variables (i.e medical history, symptoms, entry into care pathway) | baseline
  clinical variables associated with time of first doctor consultation
Socio-cognitive variables | baseline
  Socio-cognitive variables associated with time of first doctor consultation
Emotional variables | baseline
  Emotional variables associated with time of first doctor consultation
Survival | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - Centre hospitalier de Béthune, Béthune
  - Centre Hospitalier de Boulogne sur mer, Boulogne-sur-Mer
  - Centre hospitalier de Calais, Calais
  - centre Léonard de Vinci, Dechy
  - Centre d 'oncologie Dunkerquois, Dunkirk
  - CHRU, Hôpital Claude Huriez, Lille
  - Centre oscar Lambret, Lille
  - Centre hospitalier de Roubaix, Roubaix
  - Centre Hospitalier de Seclin, Seclin
  - Centre hospitalier de valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No